CLINICAL TRIAL: NCT01502787
Title: Effects of Nebivolol Versus Metoprolol on Blood Flow Responses to Exercise and Angiotensin II in Hypertensive Patients
Brief Title: Comparison of Nebivolol and Metoprolol With Exercise and Angiotensin II in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 062011-072
Record Dates: First submitted 2011-11-01; First posted 2012-01-02 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; blood pressure medications; metoprolol; nebivolol; handgrip exercise; lower body negative pressure; angiotensin II; sympathetic nerve activity; flow mediated dilation; nitric oxide; microneurography
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nebivolol; Lower Body Negative Pressure; Angiotensin II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial treatment with metoprolol (Active Comparator): The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Interventions: Drug: Metoprolol succinate; Drug: Nebivolol; Procedure: Forearm blood flow; Procedure: Microneurography; Procedure: Rhythmic handgrip exercise; Procedure: Lower body negative pressure; Drug: Angiotensin II
- Initial treatment with nebivolol (Active Comparator): The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Interventions: Drug: Metoprolol succinate; Drug: Nebivolol; Procedure: Forearm blood flow; Procedure: Microneurography; Procedure: Rhythmic handgrip exercise; Procedure: Lower body negative pressure; Drug: Angiotensin II

INTERVENTIONS:
Drug: Metoprolol succinate — The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Other Names: Toprol XL
Drug: Nebivolol — The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Other Names: Bystolic
Procedure: Forearm blood flow — Using high-resolution ultrasound, investigators will measure skeletal muscle blood flow in the forearm at rest, following handgrip exercise (described below), and following Angiotensin II infusion (described below).
Procedure: Microneurography — Investigators will measure sympathetic nerve activity from the peroneal nerve by inserting a tiny needle directly into the nerve in the leg. Investigators will localize the nerve by electrical stimulation over the skin using a blunt probe. With this stimulation, subject will notice either involuntary twitching or a tingling sensation, which may be annoying but not painful. Investigators will then introduce a tiny, sterile wire needle (an electrode) through the skin at the same location. When the tip of the needle enters the nerve, subjects may again notice involuntary muscle twitches or tingling in the leg. Investigators will then turn the electrical stimulator off and make minor adjustments in the position of the needle until investigators begin to record the nerve signals. The recording needle will remain in position throughout the study.
  Other Names: Assessment of sympathetic nerve activity (SNA)
Procedure: Rhythmic handgrip exercise — Subjects will perform a rhythmic handgrip exercise at 30% of maximal voluntary contraction for 3 minutes. Investigators will measure cardiac output (non-invasive impedance plethysmography), blood pressure, and sympathetic nerve activity (SNA) at baseline and following this handgrip exercise.
Procedure: Lower body negative pressure — Lower body negative pressure increases sympathetic nerve activity. Therefore, investigators will measure cardiac output (non-invasive impedance plethysmography), blood pressure and sympathetic nerve activity at baseline and after rhythmic handgrip exercise plus lower body negative pressure (LBNP) for 2 minutes.
  Other Names: LBNP
Drug: Angiotensin II — Investigators will measure cardiac output (non-invasive impedance plethysmography), blood pressure and sympathetic nerve activity at baseline and during intravenous infusion of Angiotensin II at the dose of 1, 2, and 3 ng/kg/min for 15 minutes at each dose.
  Other Names: IND #103,935

SUMMARY:
The purpose of this study is to determine if Nebivolol a) attenuates the angiotensin II (Ang II)-induced increase in oxidative stress, thereby attenuating Ang II-induced vasoconstriction; and b) attenuates sympathetic mediated vasoconstriction during exercise, thereby reducing functional skeletal muscle ischemia in hypertensive patients.

DETAILED DESCRIPTION:
In 40 untreated, stage I hypertensive subjects, Investigators will measure sympathetic nerve activity (microneurography); total forearm blood flow (high-resolution ultrasonography); skeletal muscle oxygenation (Near Infrared spectroscopy); plasma F2-isoprostanes; cardiac output (non-invasive impedance plethysmography); and blood pressure at baseline and after a) rhythmic handgrip exercise at 30% of maximal voluntary contraction alone for 3 minutes, b) rhythmic handgrip at the same intensity of exercise plus lower body negative pressure (LBNP) to activate sympathetic nerve activity (SNA) for 2 minutes, and c) during intravenous infusion of Angiotensin II at the dose of 1, 2, and 3 ng/kg/min for 15 minutes at each dose.

Each subject will then be randomized to receive 12 weeks of Nebivolol (Bystolic, 5-20 mg/day) or Metoprolol Succinate (Toprol XL, 100-300 mg/day), using a randomized crossover design. There will be a 2-week washout period between the two treatment periods. During drug treatment, blood pressure will be monitored every 4 weeks and the doses of Nebivolol and Metoprolol will be titrated to keep BP <140/90 mmHg. SNA, total forearm blood flow, skeletal muscle blood flow, muscle oxygenation, cardiac output, and blood pressure responses to Nebivolol will be compared to responses during Metoprolol in the same subjects.

ELIGIBILITY:
Inclusion Criteria:

* Stage I hypertension (140-159/90-99 mmHg)
* Men and women age 18-65

Exclusion Criteria:

* Congestive heart failure or coronary artery disease
* Blood pressure averaging >159/99 mmHg or resting heart rate < 55 bpm
* Serum creatinine > 1.4 mg/dL
* Asthma or chronic obstructive pulmonary diseases
* Left ventricular hypertrophy by echocardiography or ECG
* Pregnancy
* Hypersensitivity to beta blockers, microbubble contrast agents, or angiotensin
* Any history of substance abuse (other than tobacco)
* Concomitant drug treatment which raises endogenous nitric oxide levels such as nitrates or phosphodiesterase V inhibitors (Viagra, Levitra, or Cialis)
* History of symptomatic bradycardia or heart block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanpen Vongpatanasin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Rosenmeier JB, Dinenno FA, Fritzlar SJ, Joyner MJ. alpha1- and alpha2-adrenergic vasoconstriction is blunted in contracting human muscle. J Physiol. 2003 Mar 15;547(Pt 3):971-6. doi: 10.1113/jphysiol.2002.037937. Epub 2003 Feb 14. PMID 12588902
- [Background] Hansen J, Sander M, Thomas GD. Metabolic modulation of sympathetic vasoconstriction in exercising skeletal muscle. Acta Physiol Scand. 2000 Apr;168(4):489-503. doi: 10.1046/j.1365-201x.2000.00701.x. PMID 10759586
- [Background] Thomas GD, Sander M, Lau KS, Huang PL, Stull JT, Victor RG. Impaired metabolic modulation of alpha-adrenergic vasoconstriction in dystrophin-deficient skeletal muscle. Proc Natl Acad Sci U S A. 1998 Dec 8;95(25):15090-5. doi: 10.1073/pnas.95.25.15090. PMID 9844020
- [Background] Thomas GD, Zhang W, Victor RG. Impaired modulation of sympathetic vasoconstriction in contracting skeletal muscle of rats with chronic myocardial infarctions: role of oxidative stress. Circ Res. 2001 Apr 27;88(8):816-23. doi: 10.1161/hh0801.089341. PMID 11325874
- [Background] Chavoshan B, Sander M, Sybert TE, Hansen J, Victor RG, Thomas GD. Nitric oxide-dependent modulation of sympathetic neural control of oxygenation in exercising human skeletal muscle. J Physiol. 2002 Apr 1;540(Pt 1):377-86. doi: 10.1113/jphysiol.2001.013153. PMID 11927694
- [Background] Zhao W, Swanson SA, Ye J, Li X, Shelton JM, Zhang W, Thomas GD. Reactive oxygen species impair sympathetic vasoregulation in skeletal muscle in angiotensin II-dependent hypertension. Hypertension. 2006 Oct;48(4):637-43. doi: 10.1161/01.HYP.0000240347.51386.ea. Epub 2006 Aug 28. PMID 16940212
- [Background] Murphey LJ, Morrow JD, Sawathiparnich P, Williams GH, Vaughan DE, Brown NJ. Acute angiotensin II increases plasma F2-isoprostanes in salt-replete human hypertensives. Free Radic Biol Med. 2003 Oct 1;35(7):711-8. doi: 10.1016/s0891-5849(03)00395-2. PMID 14583335
- [Background] Dijkhorst-Oei LT, Stroes ES, Koomans HA, Rabelink TJ. Acute simultaneous stimulation of nitric oxide and oxygen radicals by angiotensin II in humans in vivo. J Cardiovasc Pharmacol. 1999 Mar;33(3):420-4. doi: 10.1097/00005344-199903000-00012. PMID 10069678
- [Background] Vittorio TJ, Lang CC, Katz SD, Packer M, Mancini DM, Jorde UP. Vasopressor response to angiotensin II infusion in patients with chronic heart failure receiving beta-blockers. Circulation. 2003 Jan 21;107(2):290-3. doi: 10.1161/01.cir.0000045666.04794.14. PMID 12538430
- [Background] Oelze M, Daiber A, Brandes RP, Hortmann M, Wenzel P, Hink U, Schulz E, Mollnau H, von Sandersleben A, Kleschyov AL, Mulsch A, Li H, Forstermann U, Munzel T. Nebivolol inhibits superoxide formation by NADPH oxidase and endothelial dysfunction in angiotensin II-treated rats. Hypertension. 2006 Oct;48(4):677-84. doi: 10.1161/01.HYP.0000239207.82326.29. Epub 2006 Aug 28. PMID 16940222
- [Background] Fratta Pasini A, Garbin U, Nava MC, Stranieri C, Davoli A, Sawamura T, Lo Cascio V, Cominacini L. Nebivolol decreases oxidative stress in essential hypertensive patients and increases nitric oxide by reducing its oxidative inactivation. J Hypertens. 2005 Mar;23(3):589-96. doi: 10.1097/01.hjh.0000160216.86597.ff. PMID 15716701
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Klingbeil AU, Schobel H, Langenfeld MR, Hilgers K, Schaufele T, Schmieder RE. Hyper-responsiveness to angiotensin II is related to cardiac structural adaptation in hypertensive subjects. J Hypertens. 1999 Jun;17(6):825-33. doi: 10.1097/00004872-199917060-00015. PMID 10459881
- [Background] Hopkins PN, Hunt SC, Jeunemaitre X, Smith B, Solorio D, Fisher ND, Hollenberg NK, Williams GH. Angiotensinogen genotype affects renal and adrenal responses to angiotensin II in essential hypertension. Circulation. 2002 Apr 23;105(16):1921-7. doi: 10.1161/01.cir.0000014684.75359.68. PMID 11997278
- [Background] Vuagnat A, Giacche M, Hopkins PN, Azizi M, Hunt SC, Vedie B, Corvol P, Williams GH, Jeunemaitre X. Blood pressure response to angiotensin II, low-density lipoprotein cholesterol and polymorphisms of the angiotensin II type 1 receptor gene in hypertensive sibling pairs. J Mol Med (Berl). 2001 May;79(4):175-83. doi: 10.1007/s001090100205. PMID 11409708
- [Background] Matsukawa T, Miyamoto T. Does infusion of ANG II increase muscle sympathetic nerve activity in patients with primary aldosteronism? Am J Physiol Regul Integr Comp Physiol. 2008 Jun;294(6):R1873-9. doi: 10.1152/ajpregu.00471.2007. Epub 2008 Mar 26. PMID 18367653
- [Background] Nodari S, Metra M, Dei Cas L. Beta-blocker treatment of patients with diastolic heart failure and arterial hypertension. A prospective, randomized, comparison of the long-term effects of atenolol vs. nebivolol. Eur J Heart Fail. 2003 Oct;5(5):621-7. doi: 10.1016/s1388-9842(03)00054-0. PMID 14607201
- [Background] Van Bortel LM, van Baak MA. Exercise tolerance with nebivolol and atenolol. Cardiovasc Drugs Ther. 1992 Jun;6(3):239-47. doi: 10.1007/BF00051145. PMID 1353367
- [Derived] Price A, Raheja P, Wang Z, Arbique D, Adams-Huet B, Mitchell JH, Victor RG, Thomas GD, Vongpatanasin W. Differential effects of nebivolol versus metoprolol on functional sympatholysis in hypertensive humans. Hypertension. 2013 Jun;61(6):1263-9. doi: 10.1161/HYPERTENSIONAHA.113.01302. Epub 2013 Apr 1. PMID 23547240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 subjects were screened but failed to meet inclusion criteria and were not included in treatment groups
Groups:
- Metoprolol First Then Nebivolol: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
  Metoprolol succinate: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
- Nebivolol First, Then Metoprolol: The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
Period: Overall Study
Arm/Group | Metoprolol First Then Nebivolol | Nebivolol First, Then Metoprolol
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period , there will be a 2-week washout period. Following washout, the subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Forearm Blood Flow
Time Frame: 12 weeks after each specified medication
Measure: Mean (Standard Deviation); unit: ml/min
Groups:
- First Intervention Metoprolol: 12 Weeks: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks.
- Second Intervention Nebivolol: 24 Weeks: The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks.
Arm/Group | First Intervention Metoprolol: 12 Weeks | Second Intervention Nebivolol: 24 Weeks
Number analyzed (Participants) | 21 | 21
ml/min | 96 (1) | 105 (13)

2. Secondary Outcome: Blood Pressure During Exercise
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Initial Treatment With Metoprolol | Initial Treatment With Nebivolol
Number analyzed (Participants) | 21 | 21
mmHg | 101 (3) | 103 (3)

3. Secondary Outcome: Blood Pressure During Angiotensin II Infusion
Time Frame: 12 weeks after initiation of metoprolol
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Metoprolol; Nebivolol: Angiotensin II: blood pressure was measured at baseline and during intravenous infusion of Angiotensin II at the dose of 1, 2, and 3 ng/kg/min for 15 minutes at each dose.
Arm/Group | Metoprolol | Nebivolol
Number analyzed (Participants) | 21 | 21
mmHg | 114 (3) | 113 (3)

ADVERSE EVENTS:
Groups:
- Metoprolol 21 Subjects: The subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks.
- Nebivolol 21 Subjects: The subject will be started on nebivolol (Bystolic) 5-20mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued. There will be a 2-week washout period. Following washout, the subject will be started on metoprolol succinate (Toprol XL) 100-300mg daily, which he or she will continue for a period of 12 weeks. Following the 12-week treatment period, the procedures listed below will be performed. After completion of the study procedures, the medication will be discontinued.
Arm/Group | Metoprolol 21 Subjects | Nebivolol 21 Subjects
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-07-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT01502787/Prot_SAP_000.pdf